CLINICAL TRIAL: NCT01197404
Title: Affect Management Intervention for Early Adolescents With Mental Health Problems
Brief Title: Affect Management for Early Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01NR011906 (NIH)
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: HIV Prevention
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Health Promotion (Active Comparator)
  Interventions: Behavioral: General Health Promotion
- Affect Management (Experimental)
  Interventions: Behavioral: Affect Management

INTERVENTIONS:
Behavioral: Affect Management — 12-session group intervention including affect management training as well as sexual health skills training.
  Arms: Affect Management
Behavioral: General Health Promotion — 12-session group intervention including health information on a variety of developmentally relevant health topics.
  Arms: General Health Promotion

SUMMARY:
Adolescents are at risk for HIV because of sexual and drug use behavior initiated during early adolescence, and those with mental health problems appear to be particularly susceptible. Problems with managing emotions may make it difficult for early adolescents to make good decisions about sexual and substance use behaviors. This project will develop and evaluate interventions for early adolescents with mental health issues. An intervention focused on teaching affect management skills will be compared to an intervention addressing a variety of health topics to determine which intervention best reduces risk behavior among this at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Seventh graders identified by counselors at participating public school.

Exclusion Criteria:

* Adolescent is HIV positive.
* Adolescent is developmentally delayed.
* Adolescent is pregnant.
* Adolescent has a history of sexual crime.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2009-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Adolescent-reported sexual activity | 30 Months

SECONDARY OUTCOMES:
Adolescent-reported condom use | 30 Months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Houck, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Houck CD, Hadley W, Barker D, Brown LK, Hancock E, Almy B. An Emotion Regulation Intervention to Reduce Risk Behaviors Among at-Risk Early Adolescents. Prev Sci. 2016 Jan;17(1):71-82. doi: 10.1007/s11121-015-0597-0. PMID 26297499
- [Derived] Houck CD, Barker DH, Hadley W, Menefee M, Brown LK. Sexual Risk Outcomes of an Emotion Regulation Intervention for At-Risk Early Adolescents. Pediatrics. 2018 Jun;141(6):e20172525. doi: 10.1542/peds.2017-2525. Epub 2018 May 10. PMID 29748192
- [Derived] Houck CD, Barker D, Rizzo C, Hancock E, Norton A, Brown LK. Sexting and sexual behavior in at-risk adolescents. Pediatrics. 2014 Feb;133(2):e276-82. doi: 10.1542/peds.2013-1157. Epub 2014 Jan 6. PMID 24394678